CLINICAL TRIAL: NCT05427565
Title: Exploring the Cortical Hemodynamic Variability of Four Weeks iTBS on a Healthy Participant: a Case Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Georg Kranz, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSEARS20200120005-02
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: Theta-Burst stimulation (iTBS); Functional near-infrared spectroscopy (fNIRS); Concurrent TMS/fNIRS; Prefrontal hemodynamic response; Longitudinal effects
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: One healthy participant will undergo four weeks of concurrent TBS/fNIRS to investigate the cortical hemodynamic variability
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cortical hemodynamic variability of four weeks iTBS (Experimental): One healthy participant will be included in this study, which lasts for 4 weeks, 5 visits per week, involving 20 visits in total.
  The participant will receive the following instructions the night before: to take 200 mg of caffeine one hour before the visit (no other caffeine intake since the wake-up) or avoid caffeine intake at all before the visit; to attend the visit in the morning or afternoon. These assignments will be randomized in a counterbalanced manner.
  Interventions: Other: caffeine; Other: Experimental time

INTERVENTIONS:
Other: caffeine — The investigators will ask participant to only intake 200 mg of caffeine one hour before the experiment (no other caffeine intake since the wake-up) or avoid caffeine intake at all before the experiment
Other: Experimental time — The investigators will ask participant to attend the experiment in the morning or afternoon

SUMMARY:
This study will investigate the effect of caffeine and time of day on brain excitability using excitatory brain stimulation. The investigators will recruit a healthy participant and conduct a concurrent iTBS/fNIRS protocol for 20 consecutive sessions over four weeks with or without caffeine consumption before the stimulation. Moreover, the experiment will be conducted at different times of the day (morning or afternoon)

DETAILED DESCRIPTION:
One healthy participant will be recruited for this study. The participants will be subjected to concurrent TBS/fNIRS, to which the iTBS will be applied on the left DLPFC and the NIRS will measure the prefrontal hemodynamic response simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed

Exclusion Criteria:

* history of epilepsy, seizures, or convulsions
* current or past diagnosis of neurological disorders, such as head injuries, strokes, encephalitis, epilepsy, Parkinson's, or Alzheimer's
* current or past diagnosis of psychiatric disorders, such as depression, anxiety, schizophrenia, or autism
* with metal implants, such as a cochlear implant, neurostimulator, or cardiac pacemaker

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Oxygenated hemoglobin (HbO) change compared to baseline | During and post TBS-fNIRS measurement, up to 1 month
  iTBS-induced HbO change in the DLPFC before, during and after stimulation

SECONDARY OUTCOMES:
Deoxygenated hemoglobin (HbR) change compared to baseline | During and post TBS-fNIRS measurement, up to 1 month
  iTBS-induced HbO change in the DLPFC before, during and after stimulation
Oxygen saturation change compared to baseline | During and post TBS-fNIRS measurement, up to 1 month
  iTBS-induced HbO change in the DLPFC before, during and after stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Georg S Kranz, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong